CLINICAL TRIAL: NCT04966676
Title: Beyond Chemotherapy: Nivolumab-Ipilimumab With cfDNA-guided Treatment Intensification as a Chemotherapy-sparing Strategy in Metastatic Non-small Cell Lung Cancer
Brief Title: Study of Nivolumab-Ipilimumab and cfDNA in Lung Cancer
Acronym: ATLAS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: University Health Network, Toronto (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATLAS
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Ipilimumab; CTLA-4 Antigen; Platinum Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-Small cell Lung Cancer (Experimental): Nivolumab, intravenously (given by vein), once every 3 weeks Ipilimumab, intravenously (given by vein), once every 6 weeks
  Participants will have blood samples taken for cell free deoxyribonucleic acid (cfDNA) testing.
  If there is an increasing or stable tumor cfDNA, platinum-doublet chemotherapy will be given.
  Interventions: Diagnostic Test: cfDNA blood test; Drug: Nivolumab; Drug: Ipilimumab; Combination Product: Platinum-based Chemotherapy

INTERVENTIONS:
Diagnostic Test: cfDNA blood test — Blood sample will be taken for cfDNA testing
Drug: Nivolumab — Antineoplastic agent
  Other Names: Opdivo®, BMS-936558 or MDX1106
Drug: Ipilimumab — Antineoplastic agent
  Other Names: BMS-734016, MDX010, MDX-CTLA4
Combination Product: Platinum-based Chemotherapy — May include carboplatin with gemcitabine, or paclitaxel or pemetrexed

SUMMARY:
The purpose of this research study is to look at how effective two drugs, nivolumab and ipilimumab, are for people with non-small lung cancer that has metastasized (has spread to other parts of the body) and to see what effects these drugs have on these tumors.

DETAILED DESCRIPTION:
The study will use a special blood test to evaluate the response of the cancer to treatment. This blood test will analyze tumor DNA present in the blood (deoxyribonucleic acid, molecules that contain instructions for the development and function of cells). Patients that do not have evidence of a good response using this blood test will also undergo a short course of chemotherapy in addition to nivolumab and ipilimumab.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of screening or age of consent.
* Written informed consent obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Weight ≥ 35 kg.
* Must have a life expectancy of at least 12 weeks.
* Recurrent or newly diagnosed metastatic non-small cell lung cancer
* Tumor PDL1 status <50%.
* Non-Squamous and squamous histologies are eligible
* Histologies with targetable mutations (EGFR, ALK, ROS1) are not eligible, regardless of prior treatment with tyrosine kinase inhibitors
* No prior radiation, surgery or chemotherapy is allowed for the current diagnosis of non-small cell lung cancer
* Adequate organ and marrow function

Exclusion Criteria:

* Receipt of any conventional or investigational anticancer therapy within 21 days or palliative radiotherapy within 14 days prior to the scheduled first dose of study treatment.
* Prior receipt of any immune-mediated therapy.
* Incomplete surgical resection
* Concurrent enrolment in another therapeutic clinical study. Enrolment in observational studies will be allowed.
* Any toxicity (excluding alopecia) from prior standard therapy that has not been completely resolved to baseline at the time of consent.
* Participants with prior history of myocardial infarction, transient ischemic attack, congestive heart failure ≥ Class 3 based on New York Heart Association Functional Classification or stroke within the past 3 months prior to the scheduled first dose of study treatment.
* Active or prior documented autoimmune disorders within the past 3 years prior to the scheduled first dose of study treatment with exceptions.
* Participants with confirmed human immunodeficiency virus (even if viral load is undetectable), chronic or active hepatitis B or C, or active hepatitis A.
* History of primary immunodeficiency, solid organ transplantation, or active tuberculosis (by clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice).
* Other invasive malignancy within 2 years. Non-invasive malignancies (i.e., cervical carcinoma in situ, in situ prostate cancer, non-melanomatous carcinoma of the skin, ductal carcinoma in situ of the breast that has been surgically cured) are excluded from this definition.
* Known allergy or hypersensitivity to investigational product formulations.
* History of more than one event of infusion related reactions requiring permanent discontinuation of intravenous drug treatment.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection requiring antibiotic therapy, uncontrolled hypertension, bleeding diatheses, or psychiatric illness/social situations that would limit compliance with study requirements, substantially increase risk of incurring adverse events, or compromise the ability of the subject to give written informed consent.
* Current or prior use of immunosuppressive medication within 14 days prior to the scheduled first dose of study treatment with exceptions.
* Receipt of live, attenuated vaccine within 30 days prior to the scheduled first dose of study treatment - Major surgery within 28 days prior to scheduled first dose of study treatment or still recovering from prior surgery.
* Females who are pregnant, lactating, or intend to become pregnant during their participation in the study.
* Participants who are involuntarily incarcerated or are unable to willingly provide consent or are unable to comply with the protocol procedures.
* Any condition that, in the opinion of the investigator, would interfere with safe administration or evaluation of the investigational products or interpretation of subject safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Percentage of participants whose disease does not worsen (progression-free survival rate) at 6 months | 6 months
  Progression-free survival (PFS) and 6-month PFS rate, as per RECIST 1.1, will be estimated using the Kaplan-Meier method together with their 95% confidence limit. The PFS of the study cohort will be compared to the historical controls derived from the CM9LA study.

SECONDARY OUTCOMES:
Average percentage of tumor cfDNA detected in the blood (tumor cfDNA clearance rate) at 3 weeks | 3 weeks
  To estimate the clearance of ctDNA at 3 weeks post treatment in those receiving ipilimumab-nivolumab +/- chemotherapy
Average percentage of tumor cfDNA detected in the blood (tumor cfDNA clearance rate) at 12 weeks | 12 weeks
  To estimate the clearance of ctDNA at 12 weeks post treatment in those receiving ipilimumab-nivolumab +/- chemotherapy
Number participants with adverse events | 4 years
  To evaluate the toxicity experienced by patients receiving ipilimumab-nivolumab with cfDNA-directed treatment-intensification with platinum-based chemotherapy.
Average time from the date of study enrolment until death (overall survival) | 4 years
  To evaluate the overall survival (OS) of patients receiving ipilimumab-nivolumab with cfDNA directed treatment-intensification with platinum-based chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Sacher, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada